CLINICAL TRIAL: NCT06583655
Title: A Prospective Study of Individualized Regional Node Irradiation for Sentinel Node-positive Breast Cancer Without Axillary Dissection Based on Clinical and Genomic Risk Assessment
Brief Title: Precision Regional Node Irradiation for Sentinel Node-positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, QIWEIXIANG, Deputy Chief Physician, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024（50）
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sentinel Lymph Node Dissection alone , clinical low risk group (Experimental): patients treated with surgery and Sentinel Lymph Node Dissection alone with positive lymph node metastasis.
- Sentinel Lymph Node Dissection alone , clinical high risk but genomic low risk group (Experimental): patients treated with surgery and Sentinel Lymph Node Dissection alone with positive lymph node metastasis.
- Sentinel Lymph Node Dissection alone ,clinical high risk and genomic high risk group (Experimental): patients treated with surgery and Sentinel Lymph Node Dissection alone with positive lymph node metastasis.
- with Sentinel Lymph Node Dissection(SLND) + axillary lymph node dissection(ALND) (Active Comparator): patients treated with surgery and Sentinel Lymph Node Dissection and ALND with positive lymph node metastasis.
  Interventions: Radiation: Sentinel Lymph Node Dissection(SLND) + axillary lymph node dissection(ALND)

INTERVENTIONS:
Radiation: SLND(clinical low risk) — treated with whole breast irradiation(WBI)alone 50Gy/25Fx + 10Gy/5Fx or 40Gy/15Fx + 10Gy/4Fx or no PMRT
Radiation: SLND(clinical high risk, genomic low risk) — treated with whole breast irradiation(WBI)/Post-Mastectomy Adjuvant Radiotherapy(PMRT) + regional node irradiation (Axillary +supraclavicular radiotherapy),the radiation dose could be conventional radiation or hypo-fraction irradiation:50Gy/25Fx + 10Gy/5Fx or 40Gy/15Fx + 10Gy/4Fx
Radiation: SLND alone ,clinical high risk and genomic high risk group — treated with whole breast irradiation(WBI)/Post-Mastectomy Adjuvant Radiotherapy(PMRT) + regional node irradiation (Internal Mammary Node Irradiation+ axillary +supraclavicular radiotherapy),the radiation dose could be conventional radiation or hypo-fraction irradiation:50Gy/25Fx + 10Gy/5Fx or 40Gy/15Fx + 10Gy/4Fx
Radiation: Sentinel Lymph Node Dissection(SLND) + axillary lymph node dissection(ALND) — treated with whole breast irradiation(WBI)/Post-Mastectomy Adjuvant Radiotherapy(PMRT) + regional node irradiation (Internal Mammary Node +supraclavicular radiotherapy),the radiation dose could be conventional radiation or hypo-fraction irradiation:50Gy/25Fx + 10Gy/5Fx or 40Gy/15Fx + 10Gy/4Fx
  Arms: with Sentinel Lymph Node Dissection(SLND) + axillary lymph node dissection(ALND)

SUMMARY:
Axillary lymph node dissection has long been regarded as standard if treatment of the axilla is indicated for patients with a positive sentinel node. Although axillary lymph node dissection provides excellent regional control, it is associated with harmful side-effects. Since the publication of IBCSG23-01, ACOSOG Z0011 and AMAROS study, these studies indicated that there was no significant difference in recurrence and overall survival rates between the ALNB and SLNB+ALND followed by adjuvant radiotherapy. Therefore, an adaptation of the strategy to omit axillary lymph node dissection in patients with low-risk axillary involvement who are treated with curative surgery and systematic therapy. However, they also pose new challenges for adjuvant radiotherapy decisions. In the Z0011 study, patients were required to receive breast tangent field radiotherapy. In the AMAROS study, axillary radiotherapy included level I-III axillary lymph node drainage areas and the supraclavicular area, but the study results showed a local recurrence rate of only 1.19% at 5 years in the axillary radiotherapy group. Consequently, there is considerable controversy among clinical experts about whether a combined regional lymphatic drainage area radiotherapy strategy is necessary for low-burden sentinel lymph node metastasis breast cancer patients. In contrast, results from the EORTC-22922 and MA-20 studies, which included patients undergoing axillary lymph node dissection, showed that adjuvant radiotherapy to the entire lymphatic drainage area, including the internal mammary region, reduced the risk of disease-free survival and breast cancer-specific mortality. Therefore, the adjuvant radiotherapy strategy for early breast cancer patients with low-burden sentinel lymph node metastasis remains controversial, with a lack of high-level evidence to support it.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed invasive breast cancer; 2. Age between 18 and 80 years; 3. cN0 breast cancer underwent radical surgery combined with Sentinel Lymph Node Dissection (SLND) alone with SLND positive or SLND and axillary lymph node dissection (ALND) with positive lymph node metastasis; 4. for SLND alone cohort, the regional lymph node irradiation area was determined according to the clinical risk model and genomic risk model assessment; 5. Ability to understand and willingness to participate the research and sign the consent form

Exclusion Criteria:

* • Pathologically positive ipsilateral supraclavicular lymph node

  * Pathologically or radiologically confirmed involvement of ipsilateral internal mammary lymph nodes;
  * Pregnant or lactating women;
  * Insulin dependent diabetes;
  * History of non-breast malignancy within 5 years with the exception of lobular carcinoma in situ, basal cell carcinoma of the skin, carcinoma in situ of skin and carcinoma in situ of the cervix;
  * patients have simultaneous contralateral breast cancer;
  * clinical diagnosis of distant metastatic disease;
  * Previous radiotherapy to the neck, chest and/or ipsilateral axillary region

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 205 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with arm lymphedema | 2 year
  Incidence of ipsilateral arm lymphedema 1 year after the completion of adjuvant radiotherapy

SECONDARY OUTCOMES:
Disease free survival | 5 years
  Number of patients with an oncological event (local, regional and distant recurrence free survival)
Overall survival | 5-year
  Number of patient alive after 5 years of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai jiaotong university school of medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No